CLINICAL TRIAL: NCT01761045
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Clinical Study of Monosodium L-Glutamate (MSG) and Nucleic Acid (IMP) to Evaluate the Effects on Satiety and Food Intakes at the Next Meal in Healthy Adults
Brief Title: Effect of Monosodium L-Glutamate (MSG) and Nucleic Acid (IMP) on Satiety and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AJU-S002
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Nutrition Intervention
Keywords: Monosodium L-Glutamate (MSG); Nucleic Acid (IMP); Satiety; Gastrointestinal Sensation; Consommé Soups; Snack Intake

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Soup 1 (Active Comparator): Consommé soup with Monosodium L-Glutamate (MSG)
  Interventions: Dietary Supplement: Soup 1
- Soup 2 (Active Comparator): Consommé soup with Monosodium L-Glutamate (MSG) and Nucleic Acid (IMP)
  Interventions: Dietary Supplement: Soup 2
- Soup 3 (Placebo Comparator): Placebo soup with no Monosodium L-Glutamate (MSG) or Nucleic Acid (IMP)
  Interventions: Dietary Supplement: Soup 3

INTERVENTIONS:
Dietary Supplement: Soup 1 — Consommé soup with Monosodium L-Glutamate (MSG)
  Arms: Soup 1
Dietary Supplement: Soup 2 — Consommé soup with Monosodium L-Glutamate (MSG) and Nucleic Acid (IMP)
  Arms: Soup 2
Dietary Supplement: Soup 3 — Placebo soup with no Monosodium L-Glutamate (MSG) or Nucleic Acid (IMP)
  Arms: Soup 3

SUMMARY:
The objective of this study is to confirm that Monosodium L-Glutamate (MSG) supplementation, both alone or in combination with Nucleic Acid (IMP), enhances satiety and decreases food intakes at the next meal in healthy female adults.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled, cross-over clinical trial. A total of 80 women aged 30 to 45 y will be randomized to a sequence of test product administration.

Subjects will be required to meet several inclusion and exclusion criteria, which will be assessed at the screening visit, including a general screening questionnaire, medical/medication history, eating disorder questionnaire, eating inventory questionnaire, dietary inventory questionnaire, and anthropometric and vital sign measurements. At the screening visit, a urine sample will be collected for drug and alcohol screening, cotinine level, and pregnancy. Alcohol breath test will be performed as well.

After assessment of the eligibility criteria, qualified subjects will be invited to participate in the study. This study will take approximately 3 weeks to complete.

Subjects will return to the study site within 28 days after the screening visit for testing period 1, followed by 2 additional visits (testing period 2 and 3).

Subjects will consume 1 of 3 treatments, based on randomization sequence at each test period visit: Consommé soup with Monosodium L-Glutamate (MSG), Consommé soup with MSG and Nucleic Acid (IMP), and Placebo soup with no MSG or IMP.

When subjects arrive at the research center at approximately 11:30am, admission procedures will be conducted: an alcohol breath test, food and activity diary review, and vital signs and weight will be measured. If vital sign measurements are elevated, subjects will be rescheduled within 2-3 days. Right before serving the standard lunch meal, subjects will be asked to complete a satiety motivational questionnaire. Subjects will consume the entire standard lunch meal and water within 30 min. Immediately after eating the standard lunch meal, subjects will complete the satiety motivational questionnaire.

Two hours after the standard lunch meal, subjects will be given one of the test soups (based on their randomization) to consume in its entirety, followed by completion of the satiety motivational questionnaire and the soup rating questionnaire. Fifteen minutes from test soup administration, snacks and water (ad lib) will be provided and subjects will be instructed to eat as much as or as little as they desire, followed by completing the satiety motivational questionnaire. At 3 h 15 min and at 4 h, subjects will complete the satiety motivational questionnaire.

Test periods 2 and 3 will be scheduled between 3-14 days after completing test period visit 1: all procedures are identical on each test period visit with the exception of the test treatment soup consumed by subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female, 30 to 45 yrs old
* Non-smoker
* Non-heavy Drinker
* BMI between 18.5 and 25.0 inclusive at the screening visit

Exclusion Criteria:

* History or presence of any serious and/or chronic medical or clinical disease, including renal disease, hepatic (biliary) disease, uncontrolled hypertension or uncontrolled thyroid disease, surgical conditions, cardiovascular disease other than mild hypertension or dyslipidemias, myocardial infarction, or other conditions that in the opinion of the investigator may increase the risk of participation or compromise/confound the study results
* History or diagnosis of type 1 or 2 diabetes mellitus or other uncontrolled endocrine disease
* Dysgeusia
* Any history of gastrointestinal disease or currently on treatment for a digestive disease
* Eating disorder or abnormal eating habits
* Undergone a recent significant weight change (gain or loss)
* Participating on a weight-loss program within the past 6 months prior to entry into the study
* Taking any medications for the alimentary system
* Allergy or sensitivity to foods or food additives
* History of using habitual drugs and/or alcohol abuse within the past year
* Psychosis and/or suffering from any other condition(s) which might render the individual unable to comply with the protocol or place subjects at increased risk at the discretion of the PI
* Used any investigational drug or product within the 1 month prior to the screening visit
* On special diet such as vegetarian
* Dislike the preloading soup and/or the provided lunch and/or study snacks
* Currently breast feeding and/or pregnant in the past 6 months

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Differences in food intake and subjective satiety motivational responses to treatments | 4-hr postprandial study

SECONDARY OUTCOMES:
Correlation between genetic makeup of the subject and the primary efficacy endpoints. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel S Ross, MD, Principal Investigator — The Memory Enhancement Center of America, Inc.
Locations (1):
- IBERICA Clinical Research Center, Eatontown, New Jersey, United States

REFERENCES:
- [Derived] Imada T, Hao SS, Torii K, Kimura E. Supplementing chicken broth with monosodium glutamate reduces energy intake from high fat and sweet snacks in middle-aged healthy women. Appetite. 2014 Aug;79:158-65. doi: 10.1016/j.appet.2014.04.011. Epub 2014 Apr 23. PMID 24768895